CLINICAL TRIAL: NCT04133597
Title: The Relationship Among Electroencephalography,Skin Conductance Response,Heart Rate Variability and Mental Health Among Smartphone Users After Receiving Texting or Calling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: KMUHIRB-E(I)-20170016
Record Dates: First submitted 2019-09-11; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Smartphone Users, Smartphone Addiction, Anxiety, and Skin Conductance
Keywords: skin conductance; anxiety; smartphone users; smartphone addiction
MeSH Terms: conditions — Internet Addiction Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Two experimental steps: baseline skin conductance measurements (step 1, three minutes) and measurements of SC after social media stimulation with Line messages or calls (step 2, three minutes). With a 5-minute rest period after these two steps completed, then each participant fill out questionnaires for assessing anxiety and problematic smartphone use.
  Interventions: Device: social media stimuli (Line app)

INTERVENTIONS:
Device: social media stimuli (Line app) — social media stimuli (Line app) with texting messages or calls

SUMMARY:
The number of smartphone users in Taiwan continues to increase exponentially. Smartphone addiction tends to not only disrupt the ability of social communication but cause physical and psychological problems as well. This study examined the relationship among skin conductance, electroencephalography, heart rate variability (HRV), social interaction anxiety and smartphone addiction among Line apps users, and we also tried to identify associated factors for further interventions.

ELIGIBILITY:
Inclusion Criteria:

(a) were older than 20 years of age and (b) used a smartphone with internet and Line app.

Exclusion Criteria:

the participants were those who (a) had alcoholism or drug dependence; (b) had any pre-existing major mental disorders; (c) had history of brain injury; and (d) had palmar hyperhidrosis.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
skin conductance | 3 minutes
  change of skin conductance (micro-Siemens (μS))
Heart Rate Variability (HRV) | 3 minutes
  Heart Rate Variability is a measure which indicates the variation in your heartbeats within a specific timeframe.
Electroencephalography (Hz) | 5 minutes
  Electroencephalography (EEG) is an electrophysiological monitoring method to record .... EEG is commonly recorded at sampling rates between 250 and 2000 Hz in clinical and research settings

SECONDARY OUTCOMES:
The Zung Self-Rating Anxiety Scale | 10 minutes
  The Zung Self-Rating Anxiety Scale (SAS) was developed by Zung (1971) for measuring levels of anxiety. It has been conducted in a number of cross-cultural studies, and translated into different languages with nearly 20 versions. The SAS test is a self-administered questionnaire with 20 items. The total scores of the SAS range from 20 to 80, with higher scores indicating a higher level of anxiety.
The Chinese version of Smartphone Addiction Inventory (SPAI) | 10 minutes
  The Chinese version of Smartphone Addiction Inventory (SPAI) was used to examine participant's PSU, and it was designed and developed on the basis of the Chen Internet Addiction Scale (CIAS) with a four-factor structure: compulsive behavior, functional impairment, withdrawal and tolerance [24]. The total scores of SPAI range from 26 to 104, and the higher scores indicate higher levels of smartphone addition.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No